CLINICAL TRIAL: NCT04642651
Title: Impacts of Dexmedetomidine as an Adjuvant for Femoral Nerve Block on Functional Recovery in Aged Patients After Total Knee Arthroplasty: a Randomized, Double-blinded, Controlled Trial
Brief Title: Dexmedetomidine as an Adjuvant for Femoral Nerve Block and Functional Recovery After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-502
Record Dates: First submitted 2020-11-22; First posted 2020-11-24 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Elderly; Total Knee Arthroplasty; Femoral Nerve Block; Dexmedetomidine; Functional Outcome
Keywords: Elderly; Total knee arthroplasty; Femoral nerve block; Dexmedetomidine; Functional outcome
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients in the dexmedetomidine group receive single-shot femoral nerve block preoperatively using a mixture of 0.375% ropivacaine and 1.0 μg/kg dexmedetomidine, in a total volume of 20 ml. Postoperatively, patient-controlled intravenous analgesia is provided for at least 48 hours. The formula is sufentanil (1.25 μg/ml), diluted with normal saline to 100 ml. 5-HT3 receptor antagonist is added when necessary. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients in the control group receive single-shot femoral nerve block preoperatively using a mixture of 0.375% ropivacaine and normal saline, in a total volume of 20 ml. Postoperatively, patient-controlled intravenous analgesia is provided for at least 48 hours. The formula is sufentanil (1.25 μg/ml), diluted with normal saline to 100 ml. 5-HT3 receptor antagonist is added when necessary. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in the dexmedetomidine group receive single-shot femoral nerve block preoperatively using a mixture of 0.375% ropivacaine and 1.0 μg/kg dexmedetomidine, in a total volume of 20 ml.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo — Patients in the control group receive single-shot femoral nerve block preoperatively using a mixture of 0.375% ropivacaine and normal saline, in a total volume of 20 ml.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Femoral nerve block (FNB) is a first-line analgesic technique for multimodal analgesia after total knee arthroplasty (TKA). Recent studies and meta-analysis indicate that dexmedetomidine combined with local anesthetics for FNB can prolong the analgesic duration, improve the analgesic efficacy, inhibit local inflammatory response, and reduce narcotic consumption. The investigators hypothesize that dexmedetomidine combined with ropivacaine for FNB can also improve functional recovery in aged patients after TKA.

DETAILED DESCRIPTION:
Many patients following total knee arthroplasty (TKA) complain moderate to severe postoperative pain. Multimodal analgesia, a combination of different techniques and analgesic agents, plays an increasingly important role to relieve pain after TKA. Femoral nerve block (FNB) is a first-line analgesic technique for multimodal analgesia after TKA. But local anesthetics alone often exert limited potency of analgesia and are insufficient to avoid supplemental opioid usage. Dexmedetomidine, a selective alpha 2-adrenergic receptor agonist, is widely used in clinical settings due to its properties of sedation, anxiolysis, analgesia, and sleep promotion. Recent studies and meta-analysis indicate that dexmedetomidine combined with local anesthetics for FNB can prolong the analgesic duration, improve the analgesic efficacy, inhibit local inflammatory response, and reduce narcotic consumption. The investigators hypothesize that dexmedetomidine combined with ropivacaine for FNB can also improve the functional recovery in aged patients after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years but <90 years;
* Scheduled to undergo unilateral total knee arthroplasty;
* Planned to use femoral nerve block and patient-controlled intravenous analgesia (PCIA) for multimodal analgesia.

Exclusion Criteria:

* Scheduled for bilateral total knee arthroplasty or revision surgery;
* Contraindications to femoral nerve block;
* Preoperative history of schizophrenia, myasthenia gravis, inability to communicate because of coma, severe dementia, or language barriers;
* Preoperative history of hemorrhagic disease or coagulopathy;
* Preoperative obstructive sleep apnea (diagnosed sleep apnea syndrome or a STOP-Bang score ≥3 combined with a serum bicarbonate ≥28 mmol/L);
* Sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (requirement of renal replacement therapy before surgery), or American Society of Anesthesiologists physical status >III;
* Preexistent delirium (diagnosed by Three-Dimensional Confusion Assessment Method);
* Under treatment with dexmedetomidine or clonidine.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Quality of life at 3 months after surgery-mental component summary score | At 3 months after surgery
  Quality of life is assessed with 12-item short-form (SF-12, it is summarized into physical and mental component summary scores, each ranges from 0 to 100, with higher scores indicating better quality of life).

SECONDARY OUTCOMES:
Incidence of delirium within the first 3 days after surgery | The first 3 days after surgery
  Delirium is assessed with the Three-dimensional Confusion Assessment Method (3D CAM) twice daily (8:00-10:00 and 18:00-20:00) over the first 3 postoperative hospital days. Patients with endotracheal intubation will be assessed with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) twice daily during the same period.
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of non-delirium complications (including all-cause mortality) within 30 days after surgery | Up to 30 days after surgery
  Incidence of non-delirium complications (including all-cause mortality) within 30 days after surgery
Quality of life at 3 months after surgery-physical component summary score | At 3 months after surgery
  Quality of life is assessed with 12-item short-form (SF-12, it is summarized into physical and mental component summary scores, each ranges from 0 to 100, with higher scores indicating better quality of life).
The overall subjective sleep quality at 3 months after surgery | At 3 months after surgery
  Evaluated by the Pittsburgh Sleep Quality Index, which estimates overall subjective sleep quality in the past 30 days. Overall score ranges from 0 to 21. A higher score indicates worse sleep quality, and a score greater than 5 indicates poor sleep quality.
The severity of arthritic symptoms at 3 months after surgery | At 3 months after surgery
  Assessed with WOMAC osteoarthritis index (score ranges from 0 to 96, with higher score indicating more severe symptoms).
Cognitive function at 3 months after surgery | At 3 months after surgery
  Evaluated with the modified Telephone Interview for Cognitive Status (TICS-m), a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 48, with higher score indicating better function.
Event-free survival at 3 months after surgery | At 3 months after surgery
  Time from surgery to new-onset diseases or all-cause death, whichever comes first. New-onset disease indicates those that required hospital admission and/or interventional procedure.

OTHER OUTCOMES:
Pain intensity within the first 3 days after surgery | The first 3 days after surgery
  Pain intensity is assessed twice daily (8-10 am and 18-20 pm) with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality within the first 3 days after surgery | The first 3 days after surgery
  Subjective sleep quality is assessed with the Numeric Rating Scale (NRS), an 11 points scale where 0=the best sleep and 10=the worst sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puolakka PA, Rorarius MG, Roviola M, Puolakka TJ, Nordhausen K, Lindgren L. Persistent pain following knee arthroplasty. Eur J Anaesthesiol. 2010 May;27(5):455-60. doi: 10.1097/EJA.0b013e328335b31c. PMID 20299989
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Bergeron SG, Kardash KJ, Huk OL, Zukor DJ, Antoniou J. Functional outcome of femoral versus obturator nerve block after total knee arthroplasty. Clin Orthop Relat Res. 2009 Jun;467(6):1458-62. doi: 10.1007/s11999-009-0732-y. Epub 2009 Feb 18. PMID 19224305
- [Background] Dixit V, Fathima S, Walsh SM, Seviciu A, Schwendt I, Spittler KH, Briggs D. Effectiveness of continuous versus single injection femoral nerve block for total knee arthroplasty: A double blinded, randomized trial. Knee. 2018 Aug;25(4):623-630. doi: 10.1016/j.knee.2018.04.001. Epub 2018 Apr 26. PMID 29705075
- [Background] Chan EY, Fransen M, Parker DA, Assam PN, Chua N. Femoral nerve blocks for acute postoperative pain after knee replacement surgery. Cochrane Database Syst Rev. 2014 May 13;2014(5):CD009941. doi: 10.1002/14651858.CD009941.pub2. PMID 24825360
- [Background] Mo Y, Zimmermann AE. Role of dexmedetomidine for the prevention and treatment of delirium in intensive care unit patients. Ann Pharmacother. 2013 Jun;47(6):869-76. doi: 10.1345/aph.1AR708. PMID 23719785
- [Background] Szumita PM, Baroletti SA, Anger KE, Wechsler ME. Sedation and analgesia in the intensive care unit: evaluating the role of dexmedetomidine. Am J Health Syst Pharm. 2007 Jan 1;64(1):37-44. doi: 10.2146/ajhp050508. PMID 17189578
- [Background] Arcangeli A, D'Alo C, Gaspari R. Dexmedetomidine use in general anaesthesia. Curr Drug Targets. 2009 Aug;10(8):687-95. doi: 10.2174/138945009788982423. PMID 19702517
- [Background] Peng K, Liu HY, Wu SR, Cheng H, Ji FH. Effects of Combining Dexmedetomidine and Opioids for Postoperative Intravenous Patient-controlled Analgesia: A Systematic Review and Meta-analysis. Clin J Pain. 2015 Dec;31(12):1097-104. doi: 10.1097/AJP.0000000000000219. PMID 25654534
- [Background] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534
- [Background] Deiner S, Luo X, Lin HM, Sessler DI, Saager L, Sieber FE, Lee HB, Sano M; and the Dexlirium Writing Group; Jankowski C, Bergese SD, Candiotti K, Flaherty JH, Arora H, Shander A, Rock P. Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Aug 16;152(8):e171505. doi: 10.1001/jamasurg.2017.1505. Epub 2017 Aug 16. PMID 28593326
- [Background] Wu M, Liang Y, Dai Z, Wang S. Perioperative dexmedetomidine reduces delirium after cardiac surgery: A meta-analysis of randomized controlled trials. J Clin Anesth. 2018 Nov;50:33-42. doi: 10.1016/j.jclinane.2018.06.045. Epub 2018 Jun 27. PMID 29958125
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Vorobeichik L, Brull R, Abdallah FW. Evidence basis for using perineural dexmedetomidine to enhance the quality of brachial plexus nerve blocks: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2017 Feb;118(2):167-181. doi: 10.1093/bja/aew411. PMID 28100520
- [Background] Schnabel A, Reichl SU, Weibel S, Kranke P, Zahn PK, Pogatzki-Zahn EM, Meyer-Friessem CH. Efficacy and safety of dexmedetomidine in peripheral nerve blocks: A meta-analysis and trial sequential analysis. Eur J Anaesthesiol. 2018 Oct;35(10):745-758. doi: 10.1097/EJA.0000000000000870. PMID 30095549
- [Background] Goyal R, Mittal G, Yadav AK, Sethi R, Chattopadhyay A. Adductor canal block for post-operative analgesia after simultaneous bilateral total knee replacement: A randomised controlled trial to study the effect of addition of dexmedetomidine to ropivacaine. Indian J Anaesth. 2017 Nov;61(11):903-909. doi: 10.4103/ija.IJA_277_17. PMID 29217856
- [Background] Malhotra RK, Johnstone C, Banerjee A. Dexmedetomidine in peripheral and neuraxial block: a meta-analysis. Br J Anaesth. 2014 Feb;112(2):390-1. doi: 10.1093/bja/aet568. No abstract available. PMID 24431365
- [Background] Li J, Wang H, Dong B, Ma J, Wu X. Adding dexmedetomidine to ropivacaine for femoral nerve block inhibits local inflammatory response. Minerva Anestesiol. 2017 Jun;83(6):590-597. doi: 10.23736/S0375-9393.17.11430-6. Epub 2017 Jan 20. PMID 28106354
- [Background] Packiasabapathy SK, Kashyap L, Arora MK, Batra RK, Mohan VK, Prasad G, Yadav CS. Effect of dexmedetomidine as an adjuvant to bupivacaine in femoral nerve block for perioperative analgesia in patients undergoing total knee replacement arthroplasty: A dose-response study. Saudi J Anaesth. 2017 Jul-Sep;11(3):293-298. doi: 10.4103/sja.SJA_624_16. PMID 28757829
- [Background] Wang XL, Wang J, Mu DL, Wang DX. [Dexmedetomidine combined with ropivacaine for continuous femoral nerve block improved postoperative sleep quality in elderly patients after total knee arthroplasty]. Zhonghua Yi Xue Za Zhi. 2018 Mar 13;98(10):728-732. doi: 10.3760/cma.j.issn.0376-2491.2018.10.003. Chinese. PMID 29562395
- [Background] Zhao ZF, Du L, Wang DX. Effects of dexmedetomidine as a perineural adjuvant for femoral nerve block: A systematic review and meta-analysis. PLoS One. 2020 Oct 19;15(10):e0240561. doi: 10.1371/journal.pone.0240561. eCollection 2020. PMID 33075089
- [Result] Meng ZT, Cui F, Li XY, Wang DX. Epidural morphine improves postoperative analgesia in patients after total knee arthroplasty: A randomized controlled trial. PLoS One. 2019 Jul 1;14(7):e0219116. doi: 10.1371/journal.pone.0219116. eCollection 2019. PMID 31260468